CLINICAL TRIAL: NCT01817998
Title: Role of Physical Exercise in Patients With Atrial Fibrillation.
Brief Title: Atrial Fibrillation (AF) and Physical Exercise
Acronym: EXAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Sygekassernes Helsefond (Other); Eva og Henry Frænkels Mindefond (Other); Sanofi (Industry); Thorkild Steenbecks Legat (Unknown); Toyota-Fonden (Other); Snedkermester Sophus Jacobsen and hustru Astrid Jacobsens Foundation (Other)
Responsible Party: Principal Investigator, Ane Katrine Skielboe, MD, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2-2012-048
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Intensity Endurance Physical Exercise (Experimental): High Intensity endurance physical exercise, intensity measured on Borg Scale with progression from Borg 10-13 (50% of maximum) to 17-18 (80 % of maximum). One hour of exercise twice weekly for 12 weeks supervised by physiotherapists.
  Interventions: Other: Physical Exercise
- Low Intensity Endurance Physical Exercise (Active Comparator): Low Intensity endurance physical exercise, intensity measured on Borg Scale, Borg 10-13 (50% of maximum) with no progression in intensity. One hour of exercise twice weekly for 12 weeks supervised by physiotherapists.
  Interventions: Other: Physical Exercise

INTERVENTIONS:
Other: Physical Exercise — Comparison of high versus low intensity physical exercise in patients with atrial fibrillation.

SUMMARY:
Background and study concept:

Atrial fibrillation is the new global epidemic in cardiology. With improved survival from other cardiovascular diseases and longer living in general, the incidence and prevalence of AF rise dramatically in all developed countries with an estimated life time risk of one in four for all people above the age of 40 years. Similarly in Denmark, the prevalence is estimated to almost double within 2020. It is a fatal arrhythmia with doubled mortality compared to patients with normal sinus rhythm; this primarily caused by an increased risk of stroke and heart failure. In particular stroke is a feared complication with a 70% risk of fatal outcome or lasting handicaps and immense costs for each patient as well as in terms of health costs.

Moreover, many AF patients experience a variety of symptoms and have markedly reduced quality of life. Opposed to heart failure patients and patients who have suffered from a myocardial infarction, AF patients are not offered any sort of rehabilitation when diagnosed.

Pharmacological treatment of the arrhythmia is challenging. Most often, individual and careful risk evaluation including ultrasound of the heart is obligatory to choose optimal treatment strategy and prophylactic anticoagulation. In case a new anti-arrhythmic drug is started to restore and maintain sinus rhythm, hospitalization for at least two days with heart rhythm monitoring is required to detect any possible potentially dangerous or even fatal arrhythmia as a side effect to the treatment. Additionally, the first new oral anti-arrhythmic AF drug introduced for more than twenty-five years proved to be hazardous in a high-risk AF population and is now only used with strict precautions.

To explore the role of alternative treatment strategies and to renew handling of cardiac arrhythmia, we have therefore set out to study the role of physical exercise in AF patients.

Our specific study aims are to examine:

1. The effect of physical exercise on AF burden
2. The effect of physical exercise on the risk of cardiovascular hospitalization

Method:

Our study is an interventional, randomized exercise study. 60 patients older than 18 years with ECG-documented AF will be included if written informed consent is obtained. They will be randomized 1:1 to moderate-severe (80-85% of max capacity) or low intensity (50% of max capacity) training. Exclusion criteria are language barrier, illness inherent with an expected survival shorter than a year, other reasons preventing the patient from training, revealed serious cardiac disease during pre-tests, AF ablation within one year, permanent AF.

Both groups are first participating in a nurse-led educational and care program. The program is built on two individual consultations and one team consultation with focus on education in AF.

The patients will be thoroughly examined before randomization and after ended training period with special ultrasound of the heart, ECG-monitored test of maximal oxygen uptake on ergometer bicycle, 24 hours measurement of blood pressure and pulse, and blood samples. They will all be taught to use home ECG recorders, a new handheld device. The patients will send ECG's twice daily and if the experience cardiac symptoms for 5 months (during exercise and two months after).

When randomized the patients will be divided in teams of ten and trained on separate teams, so the physiotherapist closely can guide the patients in training at the correct intensity level.

Measurements:

During and after physical exercise the burden of atrial fibrillation is measured by tele-ECG i.e. number of ECGs with atrial fibrillation divided by total number of ECGs. ECG reporting begins after four weeks of physical exercise and continues 2 months after last training session.

Recording of hospitalization begins after randomization and continues one year after last training session. All hospitalizations caused by AF or related to the AF disease (relapse of AF, heart failure, stroke, new anti-arrhythmic medication, elective electrical cardioversion, complications to anticoagulation, pacemaker implantation) are recorded. Also, total days in hospital are registered.

The AF population is growing on a global scale and the disease attracts immense interest on all international cardiology congresses. New knowledge of the effect of training for the general population as well as the effect in the setting of established disease could have paramount effect for prognosis, quality of life, and health costs as pharmacological treatment is AF still holds challenges.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal or persistent atrial fibrillation documented on ECG
* male and female of age 18 and above
* written concent

Exclusion Criteria:

* established permanent atrial fibrillation
* language barrier
* severe health conditions making physical exercise impossible or life expectancy shorter than one year
* signs of severe cardiac disease during inclusion tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in burden of atrial fibrillation at 12 weeks measured by tele-ECG i.e. number og ECGs with atrial fibrillation divided by total number of ECGs | Pre-training (baseline) and after 12 weeks of training (primary endpoint)
  Further assessments: 2 months after end of training.

SECONDARY OUTCOMES:
Change from baseline in hospitalization related to atrial fibrillation at one year after end of training measured by number of admissions/contacts registered in the patients records. | Pre-training (baseline) and one year after end of training (primary endpoint)
  Hospitalization or contact to emergency rooms registered in the patients records caused by atrial fibrillation, heart failure, stroke, atrial fibrillation, ablation, side effects to atrial fibrillation medication, and pacemaker implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Dixen, Consultant, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Department of Cardiology, Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

REFERENCES:
- [Derived] Skielboe AK, Bandholm TQ, Hakmann S, Mourier M, Kallemose T, Dixen U. Cardiovascular exercise and burden of arrhythmia in patients with atrial fibrillation - A randomized controlled trial. PLoS One. 2017 Feb 23;12(2):e0170060. doi: 10.1371/journal.pone.0170060. eCollection 2017. PMID 28231325